CLINICAL TRIAL: NCT02438995
Title: Phase I Trial of Super-Selective Intraarterial Infusion of Cetuximab (Erbitux) With or Without Radiation Therapy for the Treatment of Unresectable Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Super-Selective Intraarterial Infusion of Cetuximab (Erbitux) With or Without Radiation Therapy for the Treatment of Unresectable Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor of Neurosurgery and Otolaryngology/Head and Neck Surgery, Northwell Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-182
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma, Squamous Cell; Carcinoma, Squamous Cell of Head and Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

ARMS (2):
- Cetuximab with Radiation Therapy (Experimental): For subjects receiving radiation therapy, the treatment schedule will consist of a re-irradiation dose of approximately 70 Gy over 6-7 weeks. This experimental treatment arm will add IA Cetuximab administration every three weeks up to 2 doses to this radiation schedule.
  Interventions: Drug: Intraarterial Cetxuimab (Erbitux)
- Cetuximab Alone (Experimental): For subjects who are not candidates for re-irradiation, this experimental treatment arm will include only IA Cetuximab administration every three weeks up to 2 doses.
  Interventions: Drug: Intraarterial Cetxuimab (Erbitux)

INTERVENTIONS:
Drug: Intraarterial Cetxuimab (Erbitux) — Super-Selective Intraarterial Infusion of Cetuximab (Erbitux)

SUMMARY:
This is an open-label, non-randomized, two arm, Phase I research study of superselective intraarterial Cetuximab (Erbitux) with or without radiation therapy for treatment of recurrent unresectable squamous cell carcinoma of the head and neck (HNSCC).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of ≥18 years of age.
2. Patients with a documented diagnosis of recurrent head and neck squamous cell cancer (squamous cell carcinoma, including nasopharyngeal cancer, or adenoid cystic carcinoma).

   Patients must have at least one confirmed and evaluable tumor site.* The recurrence must have bidimensional measurements by clinical examination or CT/MRI/PET scan. A confirmed recurrence site may also be biopsy-proven
3. Tumor Recurrence which is surgically unresectable
4. Patients must have a Karnofsky performance status ≥70% (or the equivalent ECOG level of 0-2) (see Appendix Performance Status Evaluation) and an expected survival of ≥ three months.
5. Patients must have adequate hematologic reserve with WBC≥3000/mm3, absolute neutrophils ≥1500/mm3 and platelets ≥100,000/ mm3. Patients who are on Coumadin must have a platelet count of ≥150,000/ mm3
6. Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL.
7. Pre-enrollment coagulation parameters (PT and PTT) must be ≤1.5X the IUNL.
8. Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
9. Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.
10. Patients who refuse surgery.

Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
3. Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.
4. Pre-existing cardiac or respiratory disorders
5. Unrelated malignancy within 3 years
6. History of hypersensitivity reactions to other EGFR inhibitors
7. Metastatic disease
8. Less than 6 months from prior Radiation Therapy (Arm 1)
9. Previous exposure to Cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of superselective intraarterial Cetuximab. | 30 days
Descriptive frequency of subjects experiencing toxicities. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

REFERENCES:
- [Derived] Tham T, White TG, Chakraborty S, Lall RR, Ortiz R, Langer DJ, Shatzkes D, Filippi CG, Kraus D, Boockvar JA, Costantino PD. Intra-arterial cetuximab for the treatment of recurrent unresectable head and neck squamous cell carcinomadagger. J Exp Ther Oncol. 2016 Nov;11(4):293-301. PMID 27849340